CLINICAL TRIAL: NCT04111484
Title: Adrenomedullins Headache Inducing Effects on Migraine Without Patients
Brief Title: Adrenomedullin Effect on Migraine Without Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Hashmat Ghanizada, MD, MD, PhD-Fellow, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: H-18020494
Record Dates: First submitted 2019-09-26; First posted 2019-10-01 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Headache, Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Adrenomedullin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Study participants and investigator will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adrenomedullin (Active Comparator): Will received 19.9 picomol/kg/min of adrenomedullin over 20 min
  Interventions: Other: Adrenomedullin
- Saline (Placebo Comparator): Saline
  Interventions: Other: Saline

INTERVENTIONS:
Other: Adrenomedullin — Adrenomedullin is a naturally found in the human body and has strong vasoactive properties.
  Arms: Adrenomedullin
Other: Saline — Placebo
  Arms: Saline

SUMMARY:
AM is a naturally occurring peptide in the body and consists of 52 amino acids. AM belongs to the calcitonin gene-related peptide (CGRP) superfamily and has several structural, physiological and pharmacological similarities to CGRP, intermdine and amylin. In a randomized double-blind, placebo controlled cross-over design 20 migraine patients without aura recruited to receive infusion of adrenomedullin or placebo (saline).

DETAILED DESCRIPTION:
AM is a naturally occurring peptide in the body and consists of 52 amino acids. AM belongs to the calcitonin gene-related peptide (CGRP) superfamily and has several structural, physiological and pharmacological similarities to CGRP, intermdine and amylin. In a randomized double-blind, placebo controlled cross-over design 20 migraine patients without aura recruited to receive infusion of adrenomedullin or placebo (saline).

A pilot study on healthy volunteers were conducted to determine tolerable dose of adrenomedullin to the main study.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years old
* 50-100 kg
* migraine without aura according International Headache Classification Disorders 3rd edition

Exclusion Criteria:

* Tension-type headaches more than 5 days a month on average over the past year.
* All other primary headache forms.-
* Headache later than 48 hours before the start of the trial.
* Daily intake of medicines of all kinds except oral contraception.
* Taking any medicine later than 4 times the plasma half-life of that drug (on the day of the trial), except oral contraception.
* Pregnant or breastfeeding women.
* Headache on the day of the trial or later than 48 hours before the administration of the trial drug / placebo
* Migraines within 3 days before the trial date.
* Anamnestic information or clinical signs (on the day of inclusion):
* Hypertension (systolic blood pressure> 150 mmHg and / or diastolic blood pressure> 100 mmHg)
* Hypotension (systolic blood pressure <90 mm Hg and / or diastolic blood pressure <50 mmHg)
* Cardiovascular diseases of all kinds, including cerebrovascular diseases.
* Anamnestic or clinical signs of mental illness or abuse.
* Patients with glaucoma or prostate hyperplasia
* Anamnestic or clinical signs of illness of any kind that the investigating physician considers relevant for participation in the trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-28 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Migraine incidance after infusion of adrenomedullin compared to placebo | 0-12 hours
  A standard headache questionnaire will be used to register headache intensity and migraine associated symptoms.

SECONDARY OUTCOMES:
Headache intensity | 0-12 hours
  Headache intensity will be measured using Visual analogue scale (0 = no pain -10 = worst pain )
Change in puls, MAP and facial flushing | 0-90 minutes
  After infusion of adrenomedullin compared to placebo

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Headache Center, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ghanizada H, Al-Karagholi MA, Arngrim N, Morch-Rasmussen M, Walker CS, Hay DL, Ashina M. Effect of Adrenomedullin on Migraine-Like Attacks in Patients With Migraine: A Randomized Crossover Study. Neurology. 2021 May 18;96(20):e2488-e2499. doi: 10.1212/WNL.0000000000011930. Epub 2021 Apr 7. PMID 33827963